CLINICAL TRIAL: NCT06283706
Title: The Tryptophan Requirement in Healthy Adults Over 60 Years
Brief Title: The Tryptophan Requirement in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1000081113
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy Aging
Keywords: elderly; healthy; tryptophan requirement; indicator amino acid oxidation; stable isotopes
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tryptophan in Adults >60y (Experimental): Tryptophan levels, up to 7 levels, will be tested in a random order in all subjects
  Interventions: Other: Tryptophan

INTERVENTIONS:
Other: Tryptophan — There are 7 different tryptophan test levels ranging from 0.5, 2, 4, 6, 8, 10, 12 mg.kg-1.day.1

SUMMARY:
The aging population is growing rapidly. For the first time ever, Canadian seniors outnumbered young adults in 2016. Aging is associated with many physical and metabolic deteriorations including the loss of muscle mass and strength, insulin resistance, increased inflammation and oxidative stress.

The muscles of our bodies are composed of proteins and proteins are made of small building blocks called amino acids. Our bodies have the ability to make some amino acids which are called the non-essential amino acids. However, there are certain amino acids that our body's need to make protein but can only be supplied from the foods that we consume. These are called essential amino acids. Tryptophan is one of the essential amino acids that the body needs. Tryptophan is required for protein synthesis and acts as a precursor for serotonin and nicotinic acid. Therefore, there may be a need for more threonine in the diet of older adults. However, the current requirement for threonine is based on studies conducted exclusively in young adults. Thus, the purpose of this study is to find out how much tryptophan older adults need.

DETAILED DESCRIPTION:
Tryptophan is an essential amino acid and must be obtained from the diet. It is required for protein synthesis and acts as a precursor for serotonin and nicotinic acid. It is of particular importance in the diet of people who receive a large percentage of their calories from cereal grains such as maize, as it is limiting in tryptophan. Therefore, accurate knowledge of tryptophan requirement is important for dietary planning particularly for older adults. In 1998, our lab determined the tryptophan requirement in young women to be 4.01 mg/kg/day, with a safe intake at 5 mg/kg/day, using the Indicator Amino Acid Oxidation method. Since then, the investigators have determined the tryptophan requirement and safe level in healthy school-age children to be 4.7 and 6 mg/kg/day. The investigators have recently found the requirements of essential amino acids such as leucine and total sulfur amino acids in older adults and have found to be higher than young adults and a difference between the sexes. Thus, there is a need to determine the threonine requirement in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Consent provided.
* Aged 60 to 90 years old.
* In good general health as evidenced by medical history, physical health and blood draw.
* Fasting blood glucose, hemoglobin A1c (HbA1c), urea, creatinine.
* Willingness to participate in the study.
* BMI <30 kg/m2.

Exclusion Criteria:

* Presence of chronic disease and/or acute illness known to affect protein/amino acid metabolism (e.g. HIV, diabetes, taking medications known to affect protein/AA metabolism (e.g. steroids).
* Inability to tolerate the diet (i.e. allergy).
* Significant weight loss during the past month or consumption of weight reducing diets.
* Significant caffeine consumption (>2 cups per day).
* Significant consumption of alcohol (>1 drink per day i.e. 1 beer or ½ glass of wine).
* Unwilling to have blood drawn from a venous access or using a ventilated hood indirect calorimeter for the purposes of the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Determination of tryptophan requirement in adults >60 years of age. | up to 24 months
  To measure the tryptophan requirement investigators will collect breath samples from participants. From these samples, investigators will measure the amount of amino acids oxidized and how much is retained in the body when graded intakes of tryptophan are consumed by the participants consuming a controlled diet.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada